CLINICAL TRIAL: NCT07246187
Title: Comparing Haloperidol to Olanzapine in the Treatment of Suspected Cannabinoid Hyperemesis in the Emergency Department
Acronym: CH2O
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mercy Bon Secours Saint Vincent Medical Center (Other)
Responsible Party: Principal Investigator, Joseph Jabour, Dr. Joseph Jabour DO FACEP, Mercy Bon Secours Saint Vincent Medical Center
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1398377
Record Dates: First submitted 2025-11-14; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cannabinoid Hyperemesis Syndrome
MeSH Terms: conditions — Cannabinoid Hyperemesis Syndrome | interventions — Haloperidol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Haloperidol arm (Active Comparator): haloperidol
  Interventions: Drug: Haloperidol
- Olanzapine arm (Active Comparator): olanzapine
  Interventions: Drug: Olanzapine 10 milligram

INTERVENTIONS:
Drug: Olanzapine 10 milligram — olanzapine 10 mg IM
  Arms: Olanzapine arm
Drug: Haloperidol — Haloperidol 5 mg IM
  Arms: Haloperidol arm

SUMMARY:
The aim of the study is to identify which medication (haloperidol or olanzapine) is most effective in treating nausea and abdominal pain associated with cannabinoid hyperemesis using a 10-point visual analog scale with intervals of 0.5.

DETAILED DESCRIPTION:
Subjects will be weighed, have blood drawn (~20 mL, 5 teaspoons) and analyzed (CBC w/diff, CMP, lipase, quantitative hcG (if female)), urinalysis with microscopy if indicated, urine drug screen, and an ECG as part of standard routine care for such complaint in the emergency department. After consent is obtained, subjects will then be asked to rate their baseline nausea and abdominal pain on two separate 10-cm visual analog scales (VASs) [0-10, 0.5 for minor symptoms, 10 for severe symptoms].

The subjects will be pre-randomized with a computer program by an unaffiliated person to evenly distribute participants. Envelopes will be prepared by pharmacy staff with the participant number and assigned study drug, Haloperidol 5 mg or Olanzapine 10 mg, to be ready for use when a patient is enrolled. Opaque or otherwise concealed syringes will be used to maintain blinding of the administering nurse. Using a standardized order set within the EMR, subjects will be given the assigned study drug intramuscularly, and the nurse will document "CH2O study drug administered" in the electronic medical record. The subject will be monitored with five cardiac leads and pulse oximeter after receiving the study drug. While receiving intravenous crystalloid and sips of oral rehydration solution as needed, patients again will score their nausea and abdominal pain 60 minutes after medication administration, using a parallel 10-point VAS with prior score(s) visible. At 60-120 minutes after treatment, the treating physician identifies discharge readiness or, failing that, provides further orders including any rescue antiemetics (ondansetron, prochlorperazine, promethazine, or metoclopramide recommended), fluids, or imaging deemed necessary. Lastly, if appropriate, record to the nearest minute the time the patient was deemed discharge ready. After the patient's ED visit, no further collaboration will be needed from the patient. The ED chart will be reviewed to collect data including ability to tolerate liquids PO at one hour, if abdominal imaging was ordered, time of medication administration to ED discharge, admission status, need for rescue antiemetic or analgesics. The subject's information will not be used or distributed for future research studies

Subjects, all physicians, nurses, ED pharmacists, research personnel, and the investigators, including the biostatistician, will be blinded to treatment allocation until the end of the trial. In case of emergency, the unblinding will be permitted.

ELIGIBILITY:
Inclusion Criteria:

* subjects must meet ONE of the below criteria AND are a near-daily to daily user of cannabis by inhalation for greater than or equal to 6 months.

  1. Have documented previous diagnosis of cannabinoid hyperemesis, or
  2. Report (or on chart review) greater than or equal to 3 episodes of emesis in a cyclic pattern separated by greater than 1 month during the preceding 2 years, or
  3. The provider suspects cannabinoid hyperemesis as the primary or equally likely primary diagnosis.

Exclusion Criteria:

* Ineligible subjects include age less than 18 years, weight less than 50 kg, pregnancy, daily benzodiazepines use, prolonged QTc interval on the electrocardiogram (ECG), breastfeeding mothers, previously known allergy to or intolerance of either study drug, subjects taking drugs that are contraindicated with haloperidol or olanzapine, subjects with Parkison's Disease, subjects already taking haloperidol, olanzapine, or other antipsychotics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Nausea VAS scale | Change from Baseline nausea before medication administration to 60-120 minutes after medication administration
  nausea symptoms on a scale of 0-10 with 0 being no nausea and 10 being the worst nausea
vomiting | Change from Baseline vomiting before medication administration to 60-120 minutes after medication administration
  vomiting symptoms on a scale of 0-10 with 0 being no vomiting and 10 being the worst vomiting
abdominal pain | Change from Baseline abdominal pain before medication administration to 60-120 minutes after medication administration
  VAS scale abdominal pain symptoms on a scale of 0-10 with 0 being no abdominal pain and 10 being the worst abdominal pain

SECONDARY OUTCOMES:
admission versus discharge | Admission versus discharge status to be determined after the patient has been reassessed for their post medication nausea, vomiting, and abdominal pain VAS score. This occurs 60-120 minutes after study drug administration.
  admission versus discharge
Ability to tolerate PO | 60-120 minutes after medication administration
  Ability to tolerate liquids by mouth, the unit is binary, yes or no

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Saint Vincent Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No outside people will be involved, single center study